CLINICAL TRIAL: NCT05677061
Title: Clinical Evaluation on HA Coated Dynamic Hip Screws for Trochanteric Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Hospitalsenheden Vest (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-KF-298036
Record Dates: First submitted 2022-12-07; First posted 2023-01-10 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Intertrochanteric Fractures
Keywords: Stable Fractures (Evans I, II, IV)
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patient and Assessor blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA-coated (Experimental): Hydroxyapatite coating on Screw thread of DHS
  Interventions: Device: Dynamic Hip Screw with HA-coating (Hiploc)
- NON-coated (Active Comparator): No coating on Screw thread of DHS
  Interventions: Device: Dynamic Hip Screw without coating (Hiploc)

INTERVENTIONS:
Device: Dynamic Hip Screw with HA-coating (Hiploc) — During surgery for pertrochanteric hip fracture a lag screw with hydroxyapatite coating on the screw thread was used to fix the fracture
  Arms: HA-coated
Device: Dynamic Hip Screw without coating (Hiploc) — During surgery for pertrochanteric hip fracture a lag screw with no coating on the screw thread was used to fix the fracture
  Arms: NON-coated

SUMMARY:
Evaluated whether HA coated dynamic hip screws can improve fixation of the screw in trochanteric femoral fractures

DETAILED DESCRIPTION:
Randomised study to determine the effect of HA coating on the stability of dynamic Hip screws used to stabilize femoral neck fractures. Stability of the screw will be determined by RSA measurements. Additionally the fracture stability will be evaluated by RSA measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable intertrochanteric femoral fractures (Evans I, II, IV)
* able to speak Danish
* able to complete the postoperative controls
* written consent

Exclusion Criteria:

* unable to follow standard hip fracture regime
* were breastfeeding
* pregnant
* terminal disease
* in need of open fracture reduction
* in need of DHS plate with an angle different from 135 degrees
* insertion of fewer than 3 tantalum beads in the femoral head (for RSA)
* TAD >20mm in two dimensions in the first postoperative x-ray
* fracture displacement >20mm in two dimensions in the first postoperative x-ray

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Lag Screw migration measured as y-translation (mm) | 6 months PO
  Lag screw migration measured as y-translation (mm) with respect to the femoral head/neck fracture segment using marker-based radiostereometry (ModelBased RSA vs 4.2 or newer) until 6 months follow-up

SECONDARY OUTCOMES:
Lag screw migration measured as translations in mm | 6 months PO
  Lag screw migration measured as translations in mm along the three orthogonal axes (x and z) and rotations in degrees about the three orthogonal axes (x, y and z) in addition to the summed translations (total translation) and summed rotations (total rotation) with respect to the femoral head/neck fracture segment using marker-based radiostereometry (ModelBased RSA vs 4.2 or newer) until 6 months follow-up
Lag screw migration measured as rotations in degrees | 6 months PO
  Lag screw migration measured as rotations in degrees about the three orthogonal axes (x, y and z) in addition to the summed summed rotations (total rotation) with respect to the femoral head/neck fracture segment using marker-based radiostereometry (ModelBased RSA vs 4.2 or newer) until 6 months follow-up
Radiological measurements | 6 months
  TAD AP+LAT, fracture reposition AP+LAT (mm)
Clinical outcomes - HHS | 6 months PO
  Change in Harris Hip Score (HHS) measured as a scale from 0 (worst) to 100 (best) from pre-operative til 6 months postoperative
Clinical outcomes - NMS | Preoperative
  New Mobility Score measured on a scale from 0 (no mobility function) to 9 (full independent mobility function) preoperative
Clinical outcomes - Leg Lengths difference | 6 months
  Leg Length difference in cm at 6 months follow-up indicate fracture impaction
Clinical outcomes - TUG test | 6 months
  Timed Up and Go Test (TUG) at 6 months follow-up (a score less than 20 seconds indicate mobility independence)

IPD SHARING:
Plan to Share IPD: No
Not possible due til GDPR restrictions

REFERENCES:
- [Derived] Krogh AC, Thillemann JK, Hansen TB, Holck K, Kristensen MT, Palm H, Stilling M. No effect of hydroxyapatite-coated sliding hip screw threads on screw migration in the femoral head/neck of pertrochanteric fractures: a randomized controlled trial using radiostereometric analysis. J Orthop Surg Res. 2023 Sep 14;18(1):686. doi: 10.1186/s13018-023-04170-0. PMID 37710269